CLINICAL TRIAL: NCT01348555
Title: Safety, Preliminary Pharmacokinetics and Bronchodilator Properties of V0162
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00162 PI 101 1A
Record Dates: First submitted 2011-04-13; First posted 2011-05-05 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V0162 (Experimental)
  Interventions: Drug: Bronchodilatator
- Placebo (Placebo Comparator)
  Interventions: Drug: Bronchodilatator

INTERVENTIONS:
Drug: Bronchodilatator
  Arms: V0162
Drug: Bronchodilatator
  Arms: Placebo

SUMMARY:
Pulmonary administered anticholinergic agents have shown their importance in the chronic obstructive pulmonary disease (COPD) management to reduce morbidity, disability and mortality. To date, the recommended treatment of moderate to severe COPD patients consist in the combination of ß2 agonist and long acting antimuscarinic compounds. There is still a medical need in new product that could exhibit both anti-inflammatory and strong bronchodilation potency. V0162 is a compound with a potent anticholinergic activity.

Secondary PD properties of V0162 could enhance the efficacy of this antimuscarinic compound and could bring new option in the treatment of this life-threatening disease.

DETAILED DESCRIPTION:
This study has two parts. Part A will be conducted in 72 healthy volunteers. Part B will be conducted in 20 patients diagnosed with COPD.

Part A The primary objective of this part of the study is to assess the local tolerability of escalating doses of V0162 in male healthy volunteers.

Part B The primary objective of this part of the study is to assess the bronchodilator properties of V0162 at the maximal tolerated dose (determined in Part A) in COPD patients.

In addition, pharmacokinetics and vital sign including ECG will be determined.

ELIGIBILITY:
Inclusion Criteria Part A:

* Male gender
* Age between 18 to 50 years included,
* 18 ≤ Body Mass Index (BMI) < 30 kg/m²,
* Who had given their written consent for their participation in the study,
* Who, in the judgement of the Investigator, are likely to be compliant during the study,
* Registered with a social security insurance system.

Inclusion Criteria Part B:

* Aged 40 to 65 years-old,
* 18 ≤ BMI < 35 kg/m2,
* Smokers ≥ 10 packs / year,
* Moderate to severe COPD
* Registered with a social security insurance system.

Exclusion Criteria Part A:

* History of asthma or significant respiratory disorder,
* History of allergic rhinitis,
* Upper respiratory tract infection in the last month,
* Blood eosinophil count ≥ 600/μL,
* Epilepsy, narrow angle glaucoma, prostatic hypertrophy or bladder neck obstruction,
* Abnormal spirography,

Exclusion Criteria Part B:

* Respiratory tract infection in the last 6 weeks,
* Asthma or significant respiratory disorder other than COPD,
* Allergic rhinitis,
* Blood eosinophil count ≥ 600/μL,
* Epilepsy, narrow angle glaucoma, moderate to severe prostatic hypertrophy or bladder neckobstruction,
* Myocardial infarction within the previous 6 months, heart failure or serious cardiac arrhythmia,
* Moderate to severe renal impairment,
* Moderate to severe hepatic impairment
* Use of short-acting b-agonist,
* Use of anticholinergics

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To assess the local tolerability of V0162 in healthy male volunteers | change from baseline in the local tolerability over 72 h after dosing
  Monitoring of parameters of the pulmonary function: spirometry measurements. Assessment of respiratory system symptoms: using a 4-point scale and assessment of dyspnoea by VAS. Monitoring for the occurrence of AEs.
  Changes in physical examination: vital signs (blood pressure and pulse rate), holter-ECG and clinical laboratory tests (biochemistry, haematology, urinalysis).

SECONDARY OUTCOMES:
To determine the PK parameters of V0162 in healthy male volunteers | 0, 5, 15, 30, 45 min, 1, 2, 4, 8, 12, 24, 48 and 72 h after dosing
  Pharmacokinetics: evaluation of the PK parameter of V0162 (measured by area under the plasma concentration-time curve (AUC)) after oral administration and of the dose proportionality.
To assess the bronchodilator properties of V0162 in COPD | 0, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 14, 20, 24, 28 and 32 h after dosing
  Monitoring of parameters of the pulmonary function through plethysmography measurements.

CONTACTS AND LOCATIONS:
Locations (2):
- SGS, Antwerp, Belgium
- SGS Aster SAS, Paris, France

REFERENCES:
- [Derived] Devillier P, Garrigue E, D'Auzers G, Monjotin N, Similowski T, Clerc T. V0162 a new long-acting bronchodilator for treatment of chronic obstructive lung diseases: preclinical and clinical results. Respir Res. 2015 Jun 8;16(1):68. doi: 10.1186/s12931-015-0227-1. PMID 26050967